CLINICAL TRIAL: NCT00432016
Title: A Randomized, Placebo-Controlled Study to Evaluate Safety, Tolerance, Pharmacokinetics and Antiviral Activity of Amdoxovir and Zidovudine in Untreated HIV-1 Infected Subjects Currently Untreated
Brief Title: Safety, Tolerance, Pharmacokinetic and Antiviral Study of Amdoxovir in Combination With Zidovudine in Adults With HIV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RFS Pharma, LLC (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: RFS-AMDX-203; ACA-AI-001-001
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2007-05-11 (Estimated); Status verified 2007-05

CONDITIONS: HIV Infections
Keywords: HIV; pharmacokinetics; zidovudine; amdoxovir; DAPD; AMDX; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine; amdoxovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: zidovudine
Drug: amdoxovir
Procedure: pharmacokinetic sampling

SUMMARY:
The purpose of this study is to determine the short term safety, tolerance, and antiviral effect of zidovudine (AZT) and amdoxovir (AMDX, DAPD) in combination, and whether the dosage for AZT can be reduced, potentially decreasing side effects, while maintaining antiviral effects.

Study hypothesis: DADP in combination with AZT is safe and effective, and AZT dosing may be reduced, resulting in lower levels of AZT-monophosphate associated with toxicity and maintaining levels of AZT-triphosphate associated with efficacy.

DETAILED DESCRIPTION:
By 2008, market data suggest that the most commonly prescribed initial treatment regimen for HIV-1 will consist of Truvada® (FTC and tenofovir disoproxil fumarate (TDF)) and Sustiva® (efavirenz (EFV)). A newly formulated drug called Atripla™ containing all three active ingredient has now been approved by the US FDA. Therefore, second line treatments that are currently in development should provide activity against resultant mutations, primarily M184V/I (17%) and much less commonly K65R (0 to 5%), and ideally prevent or be effective against mutations that may occur during second line therapy.

The goal of our program is to identify an AZT/DAPD co-formulation with reduced resistance development and an improved safety profile for the treatment of HIV infections. DAPD has increased sensitivity to M184V/I strains and is active against thymidine analog mutations (TAMs) that may have occurred during previous antiretroviral regimens. AZT offers anti-K65R activity which is believed to be conferred by the 3'-azido moiety containing pseudo-sugar structure and base components of AZT. Hence, AZT could potentially be incorporated to prevent the emergence of the K65R mutation that could limit the long-term benefit of DAPD.

Since nucleoside reverse transcriptase inhibitors (NRTIs) require intracellular phosphorylation to form their active triphosphates, it is preferable to combine NRTIs with different critical kinases. Thymidine kinase-1 is the critical enzyme for the phosphorylation of AZT to its monophosphates. The enzyme involved in the initial phosphorylation of the active metabolite of DAPD, DXG, is guanosine kinase. Nucleotide competition studies conducted using activated human peripheral blood mononuclear (PBM) cells performed with DAPD and AZT with concentrations between 0.1-10 µM demonstrated no competitive inhibition of DXG-triphosphate formation.

The approved dose for AZT is 300 mg bid, and AZT is available as a 300 mg tablet or 100 mg capsule. A previous study in 10 HIV seropositive individuals comparing cellular AZT-mono, di- and tri-phosphate nucleotides at normal and reduced doses, 100 mg tid versus 300 mg bid, demonstrated a significant decrease in plasma AZT and intracellular AZT-monophosphate (AZT-MP) levels, (AZT-MP is associated with toxicity), without significant changes in AZT-triphosphate (AZT-TP) levels in activated PBM cells or antiviral activity. These findings on the effect of AZT dose on intracellular AZT-TP are supported by computer simulations. Maximal predicted cellular levels of AZT-MP and AZT-TP at steady-state, following 200 mg bid and 300 mg bid dosing in 3,000 simulated individuals demonstrated a high overlap between the AZT-TP histograms (> 85 %), suggesting similar efficacies for the 200 and 300 mg bid doses. The low degree of overlap between the AZT-MP histograms (< 8 %) for the two dose regimens, suggests that there may be fewer toxicities with the 200 mg bid dose, supporting our hypothesis that a zidovudine dose of 200 mg bid could reduce the AZT-MP levels without compromising the AZT-TP levels that would be obtained with a 300 mg bid dose.

This 10 day, proof of principle, pharmacokinetic study will provide important information about reduced AZT dosing to support the development of an AZT/DAPD co-formulation which may prevent the emergence of K65R mutations.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infection
* Antiretroviral therapy naïve, or if experienced, no treatment within 90 days of study screening and plan to remain off therapy for the duration of the screening and study treatment period
* HIV-1 RNA ≥ 5,000 copies/mL within 30 days of study Day 1
* CD4+ count ≥ 200 cells/mm³ within 30 days of study Day 1
* Agree to the use of two forms of adequate contraception for women, one form for men
* Estimated creatinine clearance > 80 mL/min
* Serum creatinine < 1.5 g/dL
* Able to give written informed consent prior to study start and adhere to study requirements

Exclusion Criteria:

* Active alcohol or drug use which in the opinion of the Investigator will likely compromise adherence to the study requirements
* A positive urine test for amphetamines, cocaine, and/or opioids
* Currently has any active AIDS defining illness (Category C condition according to the CDC Classification System for HIV Infection 1993)
* Any active clinically significant disease or findings during screening of medical history or physical examination that in the Investigator's opinion would compromise the outcome of the study
* Receiving oral concomitant antiviral or prophylactic drugs for opportunistic infections within 30 days prior to study entry
* Receiving concomitant treatment with nephrotoxic drugs (e.g., aminoglycosides [tobramycin, gentamicin, and amikacin], amphotericin B, vancomycin, cidofovir, foscarnet, cis-platinum, pentamidine), or competitors of renal excretion (e.g., probenecid) within 30 days of study entry
* Visual abnormalities (e.g. cataracts, macular degeneration) other than non-organic decreased visual acuity
* Receiving concomitant treatment with immunosuppressive drugs within 30 days prior to study entry
* Diabetes mellitus Type 1 or 2 which is being treated or not with any anti-diabetes agents
* Current significant gastrointestinal, renal, hepatic, bronchopulmonary, biliary, neurological, cardiovascular, oncologic, allergic, or ophthalmologic diseases including history of cataracts/lens opacities
* The following laboratory values performed within 30 days prior to study Day 1:

  * Hemoglobin < 9.0 g/dL for men; 8.0 g/dL for women
  * Platelet count < 75,000 cells per mL
  * Absolute neutrophil count < 1,000 cells per mL
  * AST, ALT, alkaline phosphatase, and amylase > 3 x ULN
  * Random or fasting glucose > 121 mg/dL
  * Serum lipase > 1.5 x ULN
  * Urinalysis ≥ 2+ proteinuria and ≥ 2 cellular casts per high powered field (HPF)
* Active acute hepatitis A and/or chronic hepatitis B or C with detectable viremia
* Subjects with clinical or laboratory evidence of significantly decreased hepatic function or decompensation, irrespective of liver enzyme levels (INR > 1.3 or albumin < 30 g/l or bilirubin > 2.5 x ULN)
* Pregnant women
* Breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2007-02; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects in each arm with Grade 3 or greater treatment emergent adverse events (AE)
Plasma Cmax, Cmin, tmax, AUC0→τ, AUC0→∞, t1/2, CL/F of DAPD and AZT in each group at Days 1 and 10
Intracellular Cmax, Cmin, tmax, AUC0→τ, AUC0→∞, and t1/2 of DXG-TP, -MP and -DP and AZT-TP, -MP, and -DP at Days 1 and 10

SECONDARY OUTCOMES:
Change in viral load (plasma HIV-1 RNA) from Baseline through Day 10
Correlate intracellular DXG-TP and AZT-TP with viral response, as measured by plasma HIV-1 RNA
Quantitate DXG, AZT, and GAZT in urine with and without DAPD
Characterize viral rebound (plasma HIV-1 RNA) following drug discontinuation for 48 hr
Measure CD4+ count changes from Baseline to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Zala, MD, Principal Investigator — Hospital Privado Modelo
Locations (1):
- Hospital Privado Modelo, Buenos Aires, Argentina

REFERENCES:
- [Background] Barry MG, Khoo SH, Veal GJ, Hoggard PG, Gibbons SE, Wilkins EG, Williams O, Breckenridge AM, Back DJ. The effect of zidovudine dose on the formation of intracellular phosphorylated metabolites. AIDS. 1996 Oct;10(12):1361-7. doi: 10.1097/00002030-199610000-00008. PMID 8902065
- [Background] Bazmi HZ, Hammond JL, Cavalcanti SC, Chu CK, Schinazi RF, Mellors JW. In vitro selection of mutations in the human immunodeficiency virus type 1 reverse transcriptase that decrease susceptibility to (-)-beta-D-dioxolane-guanosine and suppress resistance to 3'-azido-3'-deoxythymidine. Antimicrob Agents Chemother. 2000 Jul;44(7):1783-8. doi: 10.1128/AAC.44.7.1783-1788.2000. PMID 10858331
- [Background] Parikh UM, Bacheler L, Koontz D, Mellors JW. The K65R mutation in human immunodeficiency virus type 1 reverse transcriptase exhibits bidirectional phenotypic antagonism with thymidine analog mutations. J Virol. 2006 May;80(10):4971-7. doi: 10.1128/JVI.80.10.4971-4977.2006. PMID 16641288
- [Background] Thompson MA, Kessler HA, Eron JJ Jr, Jacobson JM, Adda N, Shen G, Zong J, Harris J, Moxham C, Rousseau FS; DAPD-101 Study Group. Short-term safety and pharmacodynamics of amdoxovir in HIV-infected patients. AIDS. 2005 Oct 14;19(15):1607-15. doi: 10.1097/01.aids.0000186822.68606.05. PMID 16184030
- [Derived] Murphy RL, Kivel NM, Zala C, Ochoa C, Tharnish P, Mathew J, Pascual ML, Schinazi RF. Antiviral activity and tolerability of amdoxovir with zidovudine in a randomized double-blind placebo-controlled study in HIV-1-infected individuals. Antivir Ther. 2010;15(2):185-92. doi: 10.3851/IMP1514. PMID 20386073